CLINICAL TRIAL: NCT00593424
Title: Effect of Changing the Diet to Low Fat/High Carbohydrate or High Monounsaturated Fat/Low Carbohydrate on Fasting and Post Fat Load Lipoproteins of Diabetics With Moderate Hypertriglyceridemia
Brief Title: Effect of Changing Diet on Fasting and Post Fat Load Lipoproteins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 07407
Record Dates: First submitted 2008-01-04; First posted 2008-01-15 (Estimated); Last update posted 2011-09-02 (Estimated); Status verified 2011-09

CONDITIONS: Hypertriglyceridemia; Diabetes Mellitus
MeSH Terms: conditions — Hypertriglyceridemia; Diabetes Mellitus | interventions — Diet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Low Fat/High Carbohydrate
  Interventions: Other: Low Fat/High Carbohydrate
- 2 (Active Comparator): High Monounsaturated Fat/Low Carbohydrate
  Interventions: Other: High Monounsaturated Fat/Low Carbohydrate

INTERVENTIONS:
Other: Low Fat/High Carbohydrate — Low Fat/High Carbohydrate for 6 week period
  Other Names: Diet
  Arms: 1
Other: High Monounsaturated Fat/Low Carbohydrate — High Monounsaturated Fat/Low Carbohydrate for 6 week period
  Other Names: Diet
  Arms: 2

SUMMARY:
The study examines the effect of two diets on fasting and post fat load lipoproteins of subjects with type 2 diabetes with moderate hypertriglyceridemia.

ELIGIBILITY:
Inclusion Criteria:

* Male and female,
* 18 - 75 years of age
* Type 2 diabetes
* Fasting triglycerides 300 -800mg/dL

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2002-08; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Paired t-test or Wilcoxon signed rank test will be used to evaluate the change in fasting triglycerides with the diets. | At the beginning and end of each of the two diet regimens

SECONDARY OUTCOMES:
Post-prandial lipids will be evaluated by t-test or Wilcoxon signed rank test for AUC of triglyceride and remnant lipoprotein measured by immunoseparation. | At the beginning and end of each of the two diet regimens

CONTACTS AND LOCATIONS:
Overall Officials: Debra L Simmons, M.D., Principal Investigator — UAMS/CAVHS
Locations (1):
- Central Arkansas Veterans Healthcare System, Little Rock, Arkansas, United States